CLINICAL TRIAL: NCT05513690
Title: Amnioinfusion for Intrauterine Neuroprotection: A Pilot Randomized Controlled Trial
Brief Title: Amnioinfusion for Intrauterine Neuroprotection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Foundation for Society of Maternal-Fetal Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WIHRI
Record Dates: First submitted 2022-06-17; First posted 2022-08-24 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Lactic Acidemia
Keywords: Umbilical cord gases; Neonatal neurologic morbidity; Amnioinfusion

STUDY DESIGN:
Intervention Model Description: Amnioinfusion for intrapartum risk factors for neurologic morbidity versus no amnioinfusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amnioinfusion at room temperature (intervention arm) (Experimental): Routine amnioinfusion will be administered via an intrauterine catheter inserted through the cervix. Normal saline at room temperature will be infused per hospital protocol at a rate of 600 milliliters/hour for the first hour followed by 180 milliliters/hour. A plastic applicator will be used to introduce a flexible disposable general-purpose temperature probe into the uterus. The probe will be guided to the contralateral side of the uterus from the intrauterine pressure catheter. Intrauterine temperature will then be measured by DataThermII continuous temperature monitor. This monitor has accuracy of 0.1 °C and will store temperature measurements every 10 minutes until delivery. The temperature data will be downloaded into a computer software. The DataThermII has been previously used in prior research to measure intrauterine temperature.
  Interventions: Procedure: Amnioinfusion at room temperature (intervention arm)
- Standard of care (control arm) (No Intervention): Women in this group will have the temperature probe placed and temperate measured as described in experimental arm. They will otherwise receive current standard of care (i.e. no amnioinfusion).

INTERVENTIONS:
Procedure: Amnioinfusion at room temperature (intervention arm) — Routine amnioinfusion and intrauterine temperature probe sensor
  Arms: Amnioinfusion at room temperature (intervention arm)

SUMMARY:
Hypoxic ischemic encephalopathy (HIE), a serious brain injury in infants, occurs in 2-9 per 1,000 infants after delivery. Up to 60% of infants diagnosed with HIE die and 25% of the survivors have long-term neurologic deficits. Risk factors for HIE include abnormal fetal heart tracings and intrauterine infection. Therapeutic whole-body cooling of infants with HIE is standard of care after delivery, with only 7-9 at-risk infants needing to be treated to prevent one infant from suffering long-term neurologic deficits. However, animal studies show that therapeutic cooling may be more beneficial when given in utero at the time of an insult, rather than after delivery. Though therapeutic cooling in utero has yet to be explored in humans, an established in utero fluid delivery system during labor-amnioinfusion-provides a unique opportunity for in utero intervention. We propose a pilot randomized controlled trial to test the feasibility and preliminary effects of room temperature amnioinfusion on tissue injury including HIE.

DETAILED DESCRIPTION:
Hypoxic ischemic encephalopathy (HIE), a serious brain injury in infants, occurs in 2-9 per 1,000 infants after delivery. Up to 60% of infants diagnosed with HIE die and 25% of the survivors have long-term neurologic deficits. Risk factors for HIE include abnormal fetal heart tracings and intrauterine infection. In addition, maternal fever is associated with a four to five-fold increased risk of HIE. Two phases leading to HIE are recognized: neuronal death from cellular hypoxia and further injury from exhaustion of energy stores.

Therapeutic cooling of infants with HIE provides neuroprotection by reducing metabolic demands and suppressing toxic processes. Studies show that whole-body cooling of infants reduces the risk of neurologic motor and cognitive deficits with brain imaging suggesting that human infants who are cooled earlier have a greater benefit. Moreover, animal studies show that brain cooling may be more beneficial when given in utero at the time of an insult during the first phase of cellular hypoxia, rather than after delivery. Though therapeutic cooling in utero has yet to be explored in humans, an established in utero fluid delivery system-amnioinfusion- provides a unique opportunity for in utero intervention.

Amnioinfusion (AI), the administration of fluid via an intrauterine catheter inserted through the cervix, is a common intervention during labor to improve fetal heart tracings and reduce cesarean delivery. Introduced in 1983, it used warm saline due to a theoretical concern for fetal shock from cold fluids. Subsequent studies showed no advantage of warm fluids, and fluids at room temperature (~25oC) have become standard. AI can lower in utero temperature by 1.0°C (36.4°C versus 37.4°C, P<0.01). This 1.0°C degree of cooling has been associated a 6% reduction in brain energy utilization which could be protective against neurological injury. This suggests that AI can be leveraged to lower in utero and fetal temperatures to protect against neurologic injury.

Expanding the indication for AI is a novel approach to reduce neurologic injury in utero. However, there is a gap in the acceptability and efficacy of amnioinfusion for this indication. To fill this gap, we propose a pilot randomized controlled trial to test the feasibility and effects of amnioinfusion with fluids at room temperature on infants at high risk for neurologic injury including HIE.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age >18 years old
* Singleton
* Term gestational age at time of admission (>37 weeks 0 days);

Exclusion Criteria:

* Major fetal anomaly
* Active substance or alcohol use
* Contraindications to intrauterine pressure catheter placement (e.g. placental previa, human immunodeficiency virus, Hepatitis C)
* Fetal growth restriction
* Inability to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Umbilical artery lactate | Within 15 minutes of delivery
  Cord blood lactate at the time of delivery

SECONDARY OUTCOMES:
Number of eligible patients who consent to study | Throughout study completion, an average of 1 year
  Number of patients approached and consented
Ottawa Decisional self-efficacy scale | Scale collected once from date of delivery following randomization until hospital discharge but within the first week
  The Decisional Self-Efficacy Scale measures self-confidence or belief in one's ability to make decisions, including participate in shared decision making will be compared between arms. The scale consists of 11 questions on a five-point Likert scale from 0 to 5. Scores range from 0 (not at all confident) to 100 (very confident). A score of 0 means extremely low self efficacy and a score of 100 means extremely high self efficacy.
Labour Agentry Scale | Scale collected once from date of delivery following randomization until hospital discharge but within the first week
  Labour Agentry Scale, an instrument measuring expectancies and experiences of personal control during childbirth will be compared between arms. The Labour Agentry Scale consists of 29 short affirmative statements (e.g. 'I felt confident' and 'I felt tense'). Respondents were asked to rate each statement on a seven-point Likert scale from 1 (representing rarely) to 7 (representing almost always). Possible total scores for the Labour Agentry Scale range from 29 (indicating feelings of control rarely) to 203 (reflecting feelings of control almost always).
Intrauterine temperature | 10-minute intervals from date/time of randomization until date/time of delivery, assessed only until fetus is delivered or end of second stage of labor.
  Temperature of uterus
Neonatal core temperature | Within 10 minutes of birth
  Core temperature

OTHER OUTCOMES:
Electronic fetal monitoring | 10-minute intervals from date/time of randomization until date/time of delivery, assessed only until fetus is delivered or end of second stage of labor.
  Electronic fetal monitoring recordings will be obtained with external and internal monitors, as clinically indicated. Five elements of the electronic fetal monitoring recording will be extracted using the strict and unambiguous definitions from the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) criteria and then used to categorize the electronic fetal monitoring recordings into 1 of the 3 accepted categories: I, II, or III, as well as quantitatively and semi-quantitatively. The percent of each of the five categories, individual 5 elements will be collected. This methodology has been previously validated/used and published. https://pubmed.ncbi.nlm.nih.gov/29408586/.
Montevideo units | 10-minute intervals from date/time of randomization until date/time of delivery, assessed only until fetus is delivered or end of second stage of labor.
  Calculated from intrauterine pressure catheter
Number of patients with composite and individual neonatal morbidity | Collected following delivery and/or within 6 weeks postpartum
  Neonatal death, neonatal respiratory distress syndrome, supplemental oxygen, mechanical ventilation, intubation, sepsis confirmed by culture, hypoxic-ischemic encephalopathy, seizures, Apgar score <5, and neonatal intensive care unit admission
Number of patients with composite and individual maternal morbidity | Collected following delivery and/or within 6 weeks postpartum
  Amniotic fluid embolism, acute respiratory distress syndrome, pulmonary edema, intubation, post-partum hemorrhage, blood transfusion, hysterectomy, disseminated intravascular coagulation, endometritis, chorioamnionitis, and sepsis.
Number of patients with placental pathology available | For all patients who are randomization until date/time of delivery of placenta up to 6 weeks or 36 days after delivery.
  Pathologic lesions

CONTACTS AND LOCATIONS:
Overall Officials: Brock Polnaszek, MD, Principal Investigator — Waren Alpert Medical School of Brown University, Women and Infant's Hospital
Locations (1):
- Women and Infant's Hospital of Rhode Island, Providence, Rhode Island, United States